CLINICAL TRIAL: NCT00874237
Title: Thorough QT/QTc Study of Staccato® Loxapine for Inhalation in Healthy Volunteers
Brief Title: Staccato Loxapine Thorough QT/QTc Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMDC-004-107; February 26, 2009
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Thorough QT/QTc Study
Keywords: Staccato loxapine; QT/QTc; healthy volunteers; Thorough QT/QTc study; ADASUVE; inhaled loxapine
MeSH Terms: interventions — Loxapine; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind, double dummy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment sequence ABC (Other): Treatment: A = Inhaled loxapine 10 mg, B = Placebo, C = Oral moxifloxacin 400 mg
  Interventions: Drug: Inhaled loxapine; Drug: Inhaled placebo; Drug: Oral moxifloxacin; Drug: Oral placebo
- Treatment sequence ACB (Other): Treatment: A = Inhaled loxapine 10 mg, B = Placebo, C = Oral moxifloxacin 400 mg
  Interventions: Drug: Inhaled loxapine; Drug: Inhaled placebo; Drug: Oral moxifloxacin; Drug: Oral placebo
- Treatment sequence BCA (Other): Treatment: A = Inhaled loxapine 10 mg, B = Placebo, C = Oral moxifloxacin 400 mg
  Interventions: Drug: Inhaled loxapine; Drug: Inhaled placebo; Drug: Oral moxifloxacin; Drug: Oral placebo
- Treatment sequence BAC (Other): Treatment: A = Inhaled loxapine 10 mg, B = Placebo, C = Oral moxifloxacin 400 mg
  Interventions: Drug: Inhaled loxapine; Drug: Inhaled placebo; Drug: Oral moxifloxacin; Drug: Oral placebo
- Treatment sequence CAB (Other): Treatment: A = Inhaled loxapine 10 mg, B = Placebo, C = Oral moxifloxacin 400 mg
  Interventions: Drug: Inhaled loxapine; Drug: Inhaled placebo; Drug: Oral moxifloxacin; Drug: Oral placebo
- Treatment sequence CBA (Other): Treatment: A = Inhaled loxapine 10 mg, B = Placebo, C = Oral moxifloxacin 400 mg
  Interventions: Drug: Inhaled loxapine; Drug: Inhaled placebo; Drug: Oral moxifloxacin; Drug: Oral placebo

INTERVENTIONS:
Drug: Inhaled loxapine — Inhaled Staccato Loxapine 10 mg single dose
  Other Names: ADASUVE
Drug: Inhaled placebo — Inhaled Staccato placebo single dose
Drug: Oral moxifloxacin — Oral moxifloxacin 400 mg
Drug: Oral placebo — Oral placebo similar in appearance to moxifloxacin 400 mg

SUMMARY:
The purpose of the present Phase 1 study was to assess the cardiac safety of Staccato Loxapine administered to healthy volunteers in a 3 period crossover study.

DETAILED DESCRIPTION:
Primary Objective: To assess the maximum effect of Staccato Loxapine on cardiac repolarization (QTc interval duration) at the anticipated maximum clinical dose compared to placebo in healthy volunteers.

Secondary Objective: To assess the QTc versus loxapine concentration relationship following treatment with Staccato Loxapine in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are in good general health and agree to use a medically acceptable and effective birth control method throughout the study.

Exclusion Criteria:

* Subjects who have taken prescription or nonprescription medication within 5 days of treatment,
* Subjects who have had an acute illness within the last 5 days of treatment,
* Subjects who are smokers, OR
* Subjects who have an ECG abnormality at baseline.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall R. Stoltz, MD, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit Inc., Evansville, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsDoc@alexza.com

REFERENCES:
- [Result] Spyker DA, Voloshko P, Heyman ER, Cassella JV. Loxapine delivered as a thermally generated aerosol does not prolong QTc in a thorough QT/QTc study in healthy subjects. J Clin Pharmacol. 2014 Jun;54(6):665-74. doi: 10.1002/jcph.257. Epub 2014 Jan 22. PMID 24375070

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 132 subjects were screened.
Pre-assignment Details: Of the 132 subjects who were screened for the study, 69 did not meet criteria, 5 withdrew consent, 1 no show, 9 enrollment full.
  48 (36.4%) were randomized and received at least 1 dose of study medication, and 46 completed the study
Period: Overall Study
Arm/Group | Treatment Sequence ABC | Treatment Sequence ACB | Treatment Sequence BCA | Treatment Sequence BAC | Treatment Sequence CAB | Treatment Sequence CBA
Started | 8 | 8 | 8 | 8 | 8 | 8
Completed | 8 | 7 | 7 | 8 | 8 | 8
Not Completed | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- All Subjects Treated: All 6 treatment sequences
Arm/Group | All Subjects Treated
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.854 (13.481)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Maximum Effect of ADASUVE on Cardiac Repolarization (QTc Interval Duration) at the Maximum Clinical Dose Compared to Placebo
Description: Largest of the upper CIs of the time matched differences in QTcI values between the maximum of the mean difference from baseline of the QTcI interval after time matched placebo subtraction for ADASUVE treatment at 12 prespecified post inhalation times
Time Frame: 1, 2, 5, 9, 15, 30 min, 1, 3, 6, 10 and 23 hours
Population: QT population (all patients receiving both placebo and 10 mg inhaled loxapine. LSM and CI statistics were based on the individual (within subject) corrected differences between Adasuve and placebo exposures per ICH Guideline E14 for a thorough QT study.
Measure: Least Squares Mean (95% Confidence Interval); unit: mseconds
Groups:
- Inhaled Loxapine 10 mg vs Placebo Crossover Subjects: Largest upper 95% Upper Confidence Bound (msec) for Inhaled loxapine QTcI Differences from Placebo in Change from Predose Baseline
  All upper CIs < 10 msec establishes this as a negative Thorough QT/QTc Study as defined in the ICH E14 guideline, 2005,
Arm/Group | Inhaled Loxapine 10 mg vs Placebo Crossover Subjects
Number analyzed (Participants) | 45
mseconds | 5.418 [3.083 to 7.753]

2. Secondary Outcome: Cardiac Repolarization Change (QTcI) Versus Loxapine Concentration Relationship Following Treatment With Staccato Loxapine in Healthy Volunteers.
Description: QTcI change at the median loxapine concentration (32.2 mcg/mL) based on nonlinear regression of QTcI versus log of time matched serum loxapine concentrations. This analysis looks for repolarization versus concentration relationship in a positive or negative thorough QT/QTc study result.
Time Frame: 24 hours
Population: QT + PK Population (all subjects receiving placebo and loxapine who provided QTc and pharmacokinetic data).
  LSM and CI statistics were based on the individual (within subject) corrected differences between loxapine and placebo exposures per ICH Guideline E14 for a thorough QT study.
Measure: Least Squares Mean (95% Confidence Interval); unit: mseconds
Groups:
- Inhaled Loxapine 10 mg: Largest upper 95% Upper Confidence Bound (msec) for Inhaled loxapine QTcI Differences from Placebo in Change from Predose Baseline
Arm/Group | Inhaled Loxapine 10 mg
Number analyzed (Participants) | 45
mseconds | 4.238 [2.859 to 5.617]

3. Secondary Outcome: Numbers and % of Subjects With QTcI > 450 ms
Description: Numbers and Percents of Subjects with QTcI exceeding 450 ms
Time Frame: 1, 2, 5, 9, 15, 30 min, 1, 3, 6, 10 and 23 hours
Population: QT Population (all subjects receiving placebo and inhaled loxapine and providing QT data
Measure: Count of Participants; unit: Participants
Groups:
- Inhaled Loxapine 10 mg: All subjects who received inhaled loxapine 10 mg (and oral) placebo and provided QTcI data
- Inhaled Placebo: All subjects who received inhaled (and oral) placebo and provided QTcI data
Arm/Group | Inhaled Loxapine 10 mg | Inhaled Placebo
Number analyzed (Participants) | 45 | 45
Participants | 1 | 1

4. Secondary Outcome: Numbers and % of Subjects With QTcI > 480 ms
Description: Numbers and Percents of Subjects with QTcI exceeding 480 ms
Time Frame: 1, 2, 5, 9, 15, 30 min, 1, 3, 6, 10 and 23 hours
Population: QT Population (all subjects receiving placebo and inhaled loxapine and providing QT data
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Loxapine 10 mg | Inhaled Placebo
Number analyzed (Participants) | 45 | 45
Participants | 0 | 0

5. Secondary Outcome: Numbers and % of Subjects With QTcI Change > 30 ms
Description: Numbers and Percents of Subjects with QTcI increase from baseline exceeding 30 ms
Time Frame: 1, 2, 5, 9, 15, 30 min, 1, 3, 6, 10 and 23 hours
Population: QT Population (all subjects receiving placebo and inhaled loxapine and providing QT data
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Loxapine 10 mg | Inhaled Placebo
Number analyzed (Participants) | 45 | 45
Participants | 1 | 1

6. Secondary Outcome: Numbers and % of Subjects With QTcI Change > 60 ms
Description: Numbers and Percents of Subjects with QTcI increase from baseline exceeding 60 ms
Time Frame: 1, 2, 5, 9, 15, 30 min, 1, 3, 6, 10 and 23 hours
Population: QT Population (all subjects receiving placebo and inhaled loxapine and providing QT data
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Loxapine 10 mg | Inhaled Placebo
Number analyzed (Participants) | 45 | 45
Participants | 0 | 0

7. Other Pre Specified Outcome: Maximum Effect of Moxifloxacin on Cardiac Repolarization (QTc Interval Duration) Compared to Placebo (Study Assay Sensitivity)
Description: A thorough QT/QTc study may be considered to have demonstrated assay sensitivity if 1 or more of the lower 95% CI values exceeds 5 msec ant any of the 9 predetermined time points
Time Frame: 1, 1.5, 2, 2.5, 3, 5, 8, 12, and 24 hr
Population: All subjects who completed both Inhaled placebo + oral placebo and moxifloxacin 400 mg + Inhaled placebo.
  LSM and CI statistics were based on the individual (within subject) corrected differences between moxifloxacin and placebo exposures per ICH Guideline E14 for a thorough QT study.
Measure: Least Squares Mean (95% Confidence Interval); unit: mseconds
Groups:
- Oral Moxifloxacin vs Placebo Crossover Subjects: Largest lower 95% Upper Confidence Bound (msec) for moxifloxacin QTcI Differences from Placebo in Change from Predose Baseline
  Lower CI > 5 msec at 1 or more time points establishes sensitivity of the QTc assay for the study
Arm/Group | Oral Moxifloxacin vs Placebo Crossover Subjects
Number analyzed (Participants) | 45
mseconds | 8.356 [5.825 to 10.877]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were considered treatment related from the first exposure to study treatment until 30 days after the last treatment
Description: Adverse events (AEs) were assessed predose and at 14 prespecified time points as well as whenever spontaneously reported by the subjects
Groups:
- Inhaled Loxapine 10 mg: Inhaled Staccato Loxapine 10 mg single dose Oral placebo
  Inhaled loxapine: Inhaled Staccato Loxapine 10 mg single dose
  Oral placebo: Oral placebo
- Placebo: Inhaled Staccato placebo single dose Oral placebo
  Inhaled placebo: Inhaled Staccato placebo single dose
  Oral placebo: Oral placebo
- Oral Moxifloxacin: Inhaled Staccato placebo single dose Oral moxifloxacin 400 mg
  Inhaled placebo: Inhaled Staccato placebo single dose
  Oral moxifloxacin: Oral Moxifloxacin 400 mg
Arm/Group | Inhaled Loxapine 10 mg | Placebo | Oral Moxifloxacin
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 38/47 | 19/47 | 9/47
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Loxapine 10 mg (N=47) | Placebo (N=47) | Oral Moxifloxacin (N=47)
Dysgeusia (Gastrointestinal disorders) | 9 (9) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 17 (17) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 2 (2) | 4 (4) | 2 (2)
Somnolence (Nervous system disorders) | 29 (29) | 7 (7) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2) | 1 (1)
Dermatitis, contact (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
The highest approved inhaled loxapine dose of 10 mg was studied. Supratherapeutic doses were not evaluated because of tolerability concerns in healthy subjects. The inclusion of only healthy subjects is likewise a limitation of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less